CLINICAL TRIAL: NCT04035486
Title: A Phase III, Open-label, Randomized Study of Osimertinib With or Without Platinum Plus Pemetrexed Chemo, as First-line Treatment in Patients With Epidermal Growth Factor Receptor (EGFR) Mutation Positive, Locally Advanced or Metastatic Non-small Cell Lung Cancer (FLAURA2).
Brief Title: A Study of Osimertinib With or Without Chemotherapy as 1st Line Treatment in Patients With Mutated Epidermal Growth Factor Receptor Non-Small Cell Lung Cancer (FLAURA2)
Acronym: FLAURA2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5169C00001; 2019-000650-61 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-07-29 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally; Advanced; Metastatic; Carcinoma; Non-Small Cell Lung Cancer; Osimertinib; Tagrisso
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Carcinoma | interventions — osimertinib; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Osimertinib 80mg QD (Active Comparator): Osimertinib (AZD9291) 80mg QD.
  All patients randomized into this will only receive Osimertinib 80mg.
  Dose may be reduced to allow for the management of IP related toxicity.
  Interventions: Drug: Osimertinib
- Osimertinib 80 mg QD and platinum-based chemotherapy (Experimental): Osimertinib 80 mg in combination with pemetrexed (500 mg/m2) plus cisplatin (75 mg/m2) or carboplatin (AUC5) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by Osimertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Dose may be reduced to allow for the management of IP related toxicity.
  Interventions: Drug: Pemetrexed/Carboplatin; Drug: Pemetrexed/Cisplatin

INTERVENTIONS:
Drug: Osimertinib — Drug: Osimertinib (Oral)
  Other Names:
  AZD9291
  Other Names: AZD9291
  Arms: Osimertinib 80mg QD
Drug: Pemetrexed/Carboplatin — Drug: Pemetrexed (500 mg/m2) plus carboplatin (AUC5) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by Osimertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Arms: Osimertinib 80 mg QD and platinum-based chemotherapy
Drug: Pemetrexed/Cisplatin — Drug: Pemetrexed (500 mg/m2) plus cisplatin (75 mg/m2) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by Osimertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Arms: Osimertinib 80 mg QD and platinum-based chemotherapy

SUMMARY:
The reason for the study is to find out if an experimental combination of an oral medication called osimertinib (TAGRISSO®) when used in combination with chemotherapy is more effective than giving osimertinib alone for the treatment of locally advanced or metastatic non-small cell lung cancer. Some lung cancers are due to mutations in the Deoxyribonucleic acid (DNA) which, if known, can help physicians decide the best treatment for their patients. One type of mutation can occur in the gene that produces a protein on the surface of cells called the Epidermal Growth Factor Receptor (EGFR).

Osimertinib is an Epidermal Growth Factor Receptor (EGFR) tyrosine kinase inhibitor (TKI) that targets Epidermal Growth Factor Receptor (EGFR) mutations. Unfortunately, despite the benefit observed for patients treated with osimertinib, the vast majority of cancers are expected to develop resistance to the drug over time. The exact reasons why resistance develops are not fully understood but based upon clinical research it is hoped that combining osimertinib with another type of anti-cancer therapy known as chemotherapy will delay the onset of resistance and the worsening of a patient's cancer.

In total the study aims to enroll approximately 586 patients, consisting of approximately 30 patients who will participate in a safety run-in component of the trial, and approximately 556 who will receive osimertinib alone or osimertinib in combination with chemotherapy in the main trial. In the main part of the trial there is a one in two chance of receiving osimertinib alone, and the treatment is decided at random by a computer.

The study involves a Screening Period, Treatment Period, and Follow up Period. Whilst receiving study medication, it is expected patients will attend, on average, approximately 15 visits over the first 12 months and then approximately 4 visits per year afterwards. Each visit will last about 2 to 6 hours depending on the arrangement of medical assessments by the study centre.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age; patients from Japan at least 20 years of age.
2. Pathologically confirmed non-squamous Non-Small Cell Lung Cancer (NSCLC). NSCLC of mixed histology is allowed.
3. Newly diagnosed locally advanced (clinical stage IIIB, IIIC) or metastatic Non-Small Cell Lung Cancer (NSCLC) (clinical stage IVA or IVB) or recurrent Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
4. The tumor harbors 1 of the 2 common epidermal growth factor receptor (EGFR) mutations known to be associated with Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI) sensitivity (Ex19del or L858R), either alone or in combination with other epidermal growth factor receptor (EGFR) mutations, which may include T790M.
5. Patients must have untreated advanced Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
6. WHO PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks.
7. Life expectancy >12 weeks at Day 1.
8. Willing to use contraception as appropriate during the study and for a period of time after discontinuing study treatment.

Exclusion Criteria:

1. Spinal cord compression; and unstable brain metastases, with stable brain metastases who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids can be enrolled. Patients with asymptomatic brain metastases can be eligible for inclusion if in the opinion of the Investigator immediate definitive treatment is not indicated
2. Past medical history of Interstitial Lung Disease (ILD), drug-induced Interstitial Lung Disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active Interstitial Lung Disease.
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including Hep. B, Hep. C and HIV. Screening for chronic conditions is not required. Active infection will include any patients receiving treatment for infection.
4. QT prolongation or any clinically important abnormalities in rhythm.
5. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count below the lower limit of normal (<LLN)
   * Platelet count below the LLN
   * Hemoglobin <90 g/L. The use of granulocyte colony stimulating factor support, platelet transfusion and blood transfusions to meet these criteria is not permitted.
   * ALT >2.5 x the upper limit of normal (ULN) if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
   * AST >2.5 x ULN if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
   * Total bilirubin >1.5 x ULN if no liver metastases or >3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
   * Creatinine clearance <60 mL/min calculated by Cockcroft and Gault equation or 24 hour urine collection (refer to Appendix I for appropriate calculation)
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
7. Prior treatment with any systemic anti-cancer therapy for advanced Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiation including chemotherapy, biologic therapy, immunotherapy, or any investigational drug. Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including immunotherapy, biologic therapies, investigational agents are permitted as long as treatment was completed at least 12 months prior to the development of recurrent disease.
8. Prior treatment with an Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI).
9. Major surgery within 4 weeks of the first dose of investigational product (IP). Procedures such as placement of vascular access, biopsy via mediastinoscopy or biopsy via video assisted thoracoscopic surgery are permitted.
10. Radiotherapy treatment to more than 30% of the bone marrow or( with a wide field of radiation within 4 weeks of the first dose of investigational product (IP).
11. History of hypersensitivity to active or inactive excipients of investigational product (IP) or drugs with a similar chemical structure or class to investigational product (IP).

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2026-12-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A. Jänne, MD, Principal Investigator — Dana Farber Cancer Institute, 450 Brookline Avenue, LC4114, Boston, MA 02215, USA; Kunihiko Kobayashi, MD, Principal Investigator — Department of Respiratory Medicine, Saitama Medical University International Medical Center, Saitama, Japan; David Planchard, MD, Principal Investigator — Department of Medical Oncology - Institut Gustave Roussy (IGR) - Villejuif - France
Locations (130):
- United States (22):
  - Research Site, Bellflower, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, West Hollywood, California
  - Research Site, Whittier, California
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Henderson, Nevada
  - Research Site, Albany, New York
  - Research Site, Canton, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Blacksburg, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Vancouver, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Santa Fe
- Australia (6):
  - Research Site, Camperdown
  - Research Site, Chermside
  - Research Site, Elizabeth Vale
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Melbourne
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (18):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Ostrava - Vitkovice
  - Research Site, Prague
- France (4):
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Villejuif
- India (6):
  - Research Site, Belagavi
  - Research Site, Bengaluru
  - Research Site, Gūrgaon
  - Research Site, Kolkata
  - Research Site, New Delhi
  - Research Site, Pune
- Japan (14):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Himeji-shi
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Lima
  - Research Site, San Isidro
- Philippines (6):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Legaspi
  - Research Site, Quezon City
- Russia (4):
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Saint Petersburg
  - Research Site, Syktyvkar
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Poprad
- South Africa (3):
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
  - Research Site, Rondebosch
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Maidstone
  - Research Site, Manchester
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
  For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool .
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Janne PA, Planchard D, Kobayashi K, Yang JC, Liu Y, Valdiviezo N, Kim TM, Jiang L, Kagamu H, Yanagitani N, Wang J, Biswas B, Poltoratskiy A, Neron Y, Rojas C, Koubkova L, Escriu C, Ezeife DA, Mann H, Armenteros-Monterroso E, Rukazenkov Y, Lee CK; FLAURA2 Investigators. Survival with Osimertinib plus Chemotherapy in EGFR-Mutated Advanced NSCLC. N Engl J Med. 2026 Jan 1;394(1):27-38. doi: 10.1056/NEJMoa2510308. Epub 2025 Oct 17. PMID 41104938
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Janne PA, Planchard D, Kobayashi K, Cheng Y, Lee CK, Valdiviezo N, Laktionov K, Yang TY, Yu Y, Kato T, Jiang L, Chewaskulyong B, Lucien Geater S, Maurel JM, Rojas C, Takahashi T, Havel L, Shepherd FA, Tanaka K, Ghiorghiu D, Amin NP, Armenteros-Monterroso E, Huang X, Chaudhry AA, Yang JC. CNS Efficacy of Osimertinib With or Without Chemotherapy in Epidermal Growth Factor Receptor-Mutated Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2024 Mar 1;42(7):808-820. doi: 10.1200/JCO.23.02219. Epub 2023 Dec 2. PMID 38042525
- [Derived] Planchard D, Janne PA, Cheng Y, Yang JC, Yanagitani N, Kim SW, Sugawara S, Yu Y, Fan Y, Geater SL, Laktionov K, Lee CK, Valdiviezo N, Ahmed S, Maurel JM, Andrasina I, Goldman J, Ghiorghiu D, Rukazenkov Y, Todd A, Kobayashi K; FLAURA2 Investigators. Osimertinib with or without Chemotherapy in EGFR-Mutated Advanced NSCLC. N Engl J Med. 2023 Nov 23;389(21):1935-1948. doi: 10.1056/NEJMoa2306434. Epub 2023 Nov 8. PMID 37937763
- [Derived] Planchard D, Feng PH, Karaseva N, Kim SW, Kim TM, Lee CK, Poltoratskiy A, Yanagitani N, Marshall R, Huang X, Howarth P, Janne PA, Kobayashi K. Osimertinib plus platinum-pemetrexed in newly diagnosed epidermal growth factor receptor mutation-positive advanced/metastatic non-small-cell lung cancer: safety run-in results from the FLAURA2 study. ESMO Open. 2021 Oct;6(5):100271. doi: 10.1016/j.esmoop.2021.100271. Epub 2021 Sep 17. PMID 34543864
- [Derived] White MN, Piotrowska Z, Stirling K, Liu SV, Banwait MK, Cunanan K, Sequist LV, Wakelee HA, Hausrath D, Neal JW. Combining Osimertinib With Chemotherapy in EGFR-Mutant NSCLC at Progression. Clin Lung Cancer. 2021 May;22(3):201-209. doi: 10.1016/j.cllc.2021.01.010. Epub 2021 Jan 27. PMID 33610453
- [Derived] Asahina H, Tanaka K, Morita S, Maemondo M, Seike M, Okamoto I, Oizumi S, Kagamu H, Takahashi K, Kikuchi T, Isobe T, Sugio K, Kobayashi K. A Phase II Study of Osimertinib Combined With Platinum Plus Pemetrexed in Patients With EGFR-Mutated Advanced Non-Small-cell Lung Cancer: The OPAL Study (NEJ032C/LOGIK1801). Clin Lung Cancer. 2021 Mar;22(2):147-151. doi: 10.1016/j.cllc.2020.09.023. Epub 2020 Oct 16. PMID 33199228
- See also: CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5169C00001&attachmentIdentifier=3d1bc44e-ec1e-40c6-a6ac-312b3dff8d3f&fileName=D5169C00001_Redacted_CSP.pdf&versionIdentifier=
- See also: SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5169C00001&attachmentIdentifier=57120dfa-e565-471d-8468-34b8c372e94c&fileName=D5169C00001_Redacted_SAP.pdf&versionIdentifier=
- See also: CSR_Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5169C00001&attachmentIdentifier=3bd4ded8-c239-47aa-a735-ca6f63726a3f&fileName=D5169C00001_Redcated_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 587 participants were enrolled in the study, 30 in the SRI and 557 in the Randomization component of the study. 6 participants were randomized to the Randomization component but did not receive any study treatment (2 Screen Failures, 2 Subject Decision, and 2 Deaths).
Groups:
- Safety Run-In: AZD9291 + Carboplatin + Pemetrexed: Osimertinib (AZD9291) 80 mg once daily (QD) with Carboplatin (AUC of 5 mg/mL/min [AUC5]) and Pemetrexed (500 mg/m2), both administered every 3 weeks (Q3W) for 4 cycles, followed by Osimertinib 80 mg once daily plus Pemetrexed maintenance (500 mg/m2) Q3W
- Safety Run-In: AZD9291 + Cisplatin + Pemetrexed: Osimertinib (AZD9291) 80 mg once daily (QD) with Cisplatin (75 mg/m2) and Pemetrexed (500 mg/m2), both administered every 3 weeks (Q3W) for 4 cycles, followed by Osimertinib 80 mg once daily plus Pemetrexed maintenance (500 mg/m2) Q3W
- Randomized: AZD9291 + Chemo: Osimertinib (AZD9291) 80 mg in combination with pemetrexed (500 mg/m2) plus either cisplatin (75 mg/m2) or carboplatin (AUC5) on Day 1 of 21-day cycles for 4 cycles, followed by Osimertinib (AZD9291) 80 mg QD with Pemetrexed maintenance (500 mg/m2) Q3W
- Randomized: AZD9291: Osimertinib (AZD9291) 80mg QD.
Period: Overall Study
Arm/Group | Safety Run-In: AZD9291 + Carboplatin + Pemetrexed | Safety Run-In: AZD9291 + Cisplatin + Pemetrexed | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Started | 15 | 15 | 279 | 278
Completed 4 Cycles of Carboplatin/Cisplatin Treatment (At Time of Data Cut Off (03APR2023)) | 13 | 11 | 212 | 0 (Participants in this treatment did not receive Carboplatin/Cisplatin treatment.)
Ongoing Any Study Treatment (At time of Data Cut Off (03APR2023)) | 6 | 8 | 154 | 123
Received at Least One Dose of Investigational Product (Includes Osimertinib, Cisplatin, Carboplatin, or Pemetrexed) | 15 | 15 | 276 | 275
Completed (At time of Data Cut Off (03APR2023)) | 1 | 1 | 0 | 0
Not Completed | 14 | 14 | 279 | 278
Not completed — Ongoing Study at Data Cut Off (03APR2023) | 7 | 10 | 197 | 191
Not completed — Death | 6 | 3 | 70 | 77
Not completed — Screen Failure | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 11 | 9

BASELINE CHARACTERISTICS:
Population: The Safety Run-In treatment arms are based on the Safety set, which includes all participants allocated to the safety run-in group of this study and who receive at least 1 dose of study treatment (Osimertinib, Cisplatin, Carboplatin, or Pemetrexed).
  The Randomized treatment arms are based on the Full Analysis set, which includes all participants allocated to the randomized group of this study and who were randomized to a treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-In: AZD9291 + Carboplatin + Pemetrexed | Safety Run-In: AZD9291 + Cisplatin + Pemetrexed | Randomized: AZD9291 + Chemo | Randomized: AZD9291 | Total
Number analyzed (Participants) | 15 | 15 | 279 | 278 | 587
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in Years at study entry
  Years
    Age (Years) | 62.4 (12.82) | 60.4 (8.36) | 61.0 (10.03) | 60.7 (10.57) | 60.9 (10.3)
Age, Customized [Count of Participants; unit: Participants] — Age Groups in Years at study entry
  Participants
    Age Group: <50 | 4 | 2 | 38 | 44 | 88
    Age Group: >=50-<65 | 5 | 7 | 136 | 122 | 270
    Age Group: >=65-<75 | 3 | 6 | 82 | 88 | 179
    Age Group: >=75 | 3 | 0 | 23 | 24 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 9 | 10 | 173 | 169 | 361
  Sex: Male | 6 | 5 | 106 | 109 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 39 | 29 | 68
  Ethnicity: Not Hispanic or Latino | 15 | 15 | 239 | 248 | 517
  Ethnicity: Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Race: Black or African American | 0 | 0 | 2 | 3 | 5
    Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Race: American Indian or Alaska Native | 0 | 0 | 11 | 6 | 17
    Race: Asian | 13 | 9 | 179 | 176 | 377
    Race: White | 2 | 6 | 74 | 83 | 165
    Race: Other | 0 | 0 | 13 | 10 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnic population
  Participants
    Ethnic Population: Asian, not specified | 9 | 7 | 108 | 107 | 231
    Ethnic Population: Chinese | 4 | 2 | 71 | 69 | 146
    Ethnic Population: Other ethnic population (Non-Asian) | 2 | 6 | 99 | 100 | 207
    Ethnic Population: Missing | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Graded by Common Terminology Criteria for Adverse Event v5 (Safety Run-In Treatment Arms Only)
Description: Adverse events were summarized by maximum reported Common Terminology Criteria for Adverse Event (CTCAE) grade, version 5.0.
  Grade 1 (Mild): asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 (Moderate): minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 (Severe or medically significant but not immediately life-threatening): hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living.
  Grade 4 (Life-threatening consequences): urgent intervention indicated.
  Grade 5: Death related to AE.
  Includes adverse events with onset date on or after the date of first dose and up to and including 28 days following discontinuation of treatment but prior to the start of a new anti-cancer therapy.
Time Frame: From first dose date to 28 days following last dose, up to 45 months
Population: Participants from the Safety Analysis Set, which includes all participants in the Safety Run-In Treatment Arms who received at least 1 dose of study treatment (osimertinib, cisplatin, carboplatin, or pemetrexed).
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In: AZD9291 + Carboplatin + Pemetrexed | Safety Run-In: AZD9291 + Cisplatin + Pemetrexed
Number analyzed (Participants) | 15 | 15
Participants
  Grade 1 | 1 | 0
  Grade 2 | 9 | 4
  Grade 3 | 3 | 8
  Grade 4 | 0 | 2
  Grade 5 | 2 | 0
  No Adverse Events Reported | 0 | 1

2. Primary Outcome: Progression-free Survival (PFS) (Randomized Component)
Description: Progression-free survival (PFS) using Investigator assessment as defined by RECIST 1.1. Median progression free survival (months) calculated using the Kaplan-Meier method.
  Progression-free survival (PFS) is defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
  The primary efficacy analysis of the investigator-assessed progression-free survival will be performed when approximately 278 PFS events and at least 16 months of follow-up after Last subject in, has occurred in the 556 randomized patients.
Time Frame: Up to approximately 33 months after the first patient is randomized (maximum follow up of 33.3 months)
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months | 25.5 [24.7 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 16.7 [14.1 to 21.3]
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; The analysis was performed using a log rank test stratified by race (Chinese/Asian vs. Non-Chinese/Asian vs. Non-Asian), WHO performance status (0 vs. 1), and method used for tissue testing (central vs. local); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.49 to 0.79] — A hazard ratio of less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

3. Primary Outcome: Sensitivity Analysis for Progression-free Survival (PFS) by Blinded Independent Central Review (BICR) Assessment (Randomized Component)
Description: Sensitivity analysis for progression-free survival (PFS) by blinded independent central review (BICR) using Investigator assessment as defined by RECIST 1.1. Median progression free survival (months) calculated using the Kaplan-Meier method.
  Progression-free survival (PFS) is defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
  The primary efficacy analysis of the investigator-assessed progression-free survival will be performed when approximately 278 PFS events and at least 16 months of follow-up after Last subject in, has occurred in the 556 randomized patients.
Time Frame: Up to approximately 33 months after the first patient is randomized (maximum follow up of 33.2 months).
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months | 29.4 [25.1 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 19.9 [16.6 to 25.3]
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.48 to 0.80] — A hazard ratio of less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

4. Secondary Outcome: Overall Survival (OS) (Safety Run-In Treatment Arms Only)
Description: Overall survival is defined as the time from the date of first dose until death due to any causes. Subjects not known to have died at the time of analysis are censored at the last recorded date on which the subject was known to be alive. Median overall survival calculated using the Kaplan-Meier method.
  Per the protocol, the safety run-in treatment arms were combined and analyzed regardless of chemotherapy received for consistency with the randomized component.
Time Frame: Up to 45 months (maximum follow up 44.6 months)
Population: Safety Analysis Set, includes all participants in the Safety Run-In Treatment Arms who received at least 1 dose of study treatment (osimertinib, cisplatin, carboplatin, or pemetrexed).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Overall Safety Run-In Participants: Includes all participants in both Safety Run-In treatment arms: AZD9291 + Carboplatin + Pemetrexed and AZD9291 + Cisplatin + Pemetrexed
Arm/Group | Overall Safety Run-In Participants
Number analyzed (Participants) | 30
Months | NA [34.0 to NA] — Median and Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.

5. Secondary Outcome: Duration of Response (DoR) (Safety Run-In Treatment Arms Only)
Description: Duration of response (DoR) is defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression (i.e. date of progression free survival event or censoring - date of first response + 1). The end of response should coincide with the date of progression or death from any cause used for the progression free survival endpoint. The time of the initial response is defined as the latest of the dates contributing towards the first visit that was Complete response or Partial response that was subsequently confirmed.
  Per the protocol, the safety run-in treatment arms were combined and analyzed regardless of chemotherapy received for consistency with the randomized component.
Time Frame: Up to 45 months
Population: Participants from the Safety Analysis Set, which includes all participants in the Safety Run-In Treatment Arms who received at least 1 dose of study treatment (osimertinib, cisplatin, carboplatin, or pemetrexed), that had a confirmed response.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Overall Safety Run-In Participants
Number analyzed (Participants) | 26
Months | 27.5 (13.48)

6. Secondary Outcome: Objective Response Rate (ORR) (Safety Run-In Treatment Arms Only)
Description: Confirmed objective response rate (per RECIST 1.1 using Investigator assessments) is defined as the number (%) of subjects with at least 1 visit response of Completed Response (CR) or Partial Response (PR), where each CR or PR must be subsequently confirmed at least 4 weeks after the visit when the response was first observed with no evidence of progression between the initial and CR/PR confirmation visit.
  Confidence Interval is calculated using the exact Clopper-Pearson method.
  Per the protocol, the safety run-in treatment arms were combined and analyzed regardless of chemotherapy received for consistency with the randomized component.
Time Frame: Up to 45 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Overall Safety Run-In Participants
Number analyzed (Participants) | 30
Percent of Participants | 86.7 [69.28 to 96.24]

7. Secondary Outcome: Depth of Response (Percent Change From Baseline in Tumor Diameter) (Safety Run-In Treatment Arms Only)
Description: Depth of Response (percent change from Baseline in tumor diameter) is defined as the relative percent change in the sum of the longest diameters of RECIST 1.1 target lesions (TL) at the nadir in the absence of new lesions or progression of non-target lesions (NTL) compared to baseline. The best percentage change in TL size is the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction. Tumor assessments of the chest and abdomen (including the entire liver and both adrenal glands) were performed using RECIST 1.1 by the investigator on images from CT (preferred) or MRI with IV contrast.
  Per the protocol, the safety run-in treatment arms were combined and analyzed regardless of chemotherapy received for consistency with the randomized component.
Time Frame: Up to 45 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Overall Safety Run-In Participants
Number analyzed (Participants) | 30
Percent change from baseline | -57.72 (22.090)

8. Secondary Outcome: Disease Control Rate (DCR) by Investigator (Safety Run-In Treatment Arms Only)
Description: Disease control rate is defined as the percentage of subjects who have a best overall response of Complete response (CR) or Partial response (PR) or Stable disease (SD) by RECIST 1.1 as assessed by the Investigator. For participants with a best overall response of SD, a RECIST assessment of SD must have been observed at least 6 weeks minus 1 week (at least 35 study days) following the first dose.
  Per the protocol, the safety run-in treatment arms were combined and analyzed regardless of chemotherapy received for consistency with the randomized component.
Time Frame: Up to 45 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Safety Run-In Participants
Number analyzed (Participants) | 30
Participants
  Complete Response (CR) | 3
  Partial Response (PR) | 23
  Stable Disease (SD) | 4
Statistical Analysis 1: Comparison: Overall Safety Run-In Participants; A 95% CI was calculated on the percentage of participants with a Response or Stable Disease using the exact (Clopper-Pearson) method; Test type: Other; Clopper-Pearson; Percentage of Participants = 100.00, 95% CI 2-sided [88.43 to 100.00]

9. Secondary Outcome: Overall Survival (OS) (Randomized Component)
Description: Overall survival is defined as the time from the date of randomization until death due to any cause. Subjects not known to have died at the time of analysis are censored at the last recorded date on which the subject was known to be alive. Median overall Survival calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized (maximum follow up of 34.1 months)
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months | NA [31.9 to NA] — Median and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | NA [NA to NA] — Median, Lower Limit and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5238, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.65 to 1.24] — A hazard ratio of less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm; An adjusted CI of (0.54, 1.51) was computed at the 2-sided 99.84% level, considering a 2-sided significance level of 0.00158 for the overall survival interim analysis, based on the O'Brien and Fleming spending function, assuming 334 deaths for the final overall survival analysis

10. Secondary Outcome: Landmark Overall Survival (LOS) at 1, 2, and 3 Years (Randomized Component)
Description: Landmark Overall Survival at 1, 2, and 3 years looks at the percent of patients alive at 1, 2 and 3 year time points.
  Overall survival at 36 months not included to data cut off prior to 36-month timepoint.
  Overall survival percentage calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized (maximum follow up of 34.1 months)
Population: Full Analysis Set, includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
percent of participants
  Overall survival at 12 months (%) | 88.8 [84.4 to 92.0] | 92.0 [88.1 to 94.7]
  Overall survival at 24 months (%) | 78.9 [73.4 to 83.4] | 73.0 [66.9 to 78.1]

11. Secondary Outcome: Objective Response Rate (ORR) (Randomized Component)
Description: Objective Response Rate (ORR) (per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments) is defined as the number (%) of patients with at least 1 visit response of Complete Response or Partial Response. Data obtained up until progression, or the last evaluable assessment in the absence of progression, was included in the assessment of Objective Response Rate.
  The investigator-assessed ORR was summarized with a logistic regression stratified by race (Chinese/Asian vs. Non-Chinese/Asian vs. Non-Asian), WHO performance status (0 vs. 1), and method used for tissue testing (central vs. local).
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Percent of Participants | 84.40 [79.51 to 88.30] | 77.10 [71.52 to 81.85]
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; The analysis was performed using a logistic regression stratified by race (Chinese/Asian vs. Non-Chinese/Asian vs. Non-Asian), WHO performance status (0 vs. 1), and method used for tissue testing (central vs. local); Test type: Superiority; p = 0.0261, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.06 to 2.44] — And odds ratio of greater than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

12. Secondary Outcome: Duration of Response (DoR) (Randomized Component)
Description: The duration of response is defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression. The end of response should coincide with the date of progression or death from any cause used for the progression-free survival endpoint. The time of the initial response is defined as the latest of the dates contributing towards the first response of Partial response or Complete response.
  Median values of the duration of response, along with two-sided 95% CI in each treatment group were computed using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Participants from the Full Analysis Set, which includes all randomized participants, that had a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 232 | 210
Months | 24.0 [20.9 to 27.8] | 15.3 [12.7 to 19.4]

13. Secondary Outcome: Depth of Response (Percent Change From Baseline in Tumor Diameter) (Randomized Component)
Description: Depth of Response (percent change from Baseline in tumor diameter) is defined as the relative percent change in the sum of the longest diameters of RECIST 1.1 target lesions (TL) at the nadir in the absence of new lesions or progression of non-target lesions (NTL) compared to baseline. The best percentage change in TL size is the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction. Tumor assessments of the chest and abdomen (including the entire liver and both adrenal glands) were performed using RECIST 1.1 by the investigator on images from CT (preferred) or MRI with IV contrast.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 275 | 276
Percent change from baseline | -50.77 [-53.75 to -47.78] | -47.41 [-50.39 to -44.43]
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; The analysis was performed using analysis of covariance with baseline tumor size and time from baseline scan to randomization as covariates and with factors race (Chinese/Asian vs. Non-Chinese/Asian vs. Non-Asian), WHO performance status (0 vs. 1), and method used for tissue testing (central vs. local); Test type: Superiority; p = 0.1067, ANCOVA; Least Square Mean Difference = -3.36, 95% CI 2-sided [-7.44 to 0.72] — A difference in least square means less than 0 favors the Osimertinib (AZD9291) + Chemo treatment arm

14. Secondary Outcome: Disease Control Rate (DCR) by Investigator (Randomized Component)
Description: Disease control rate (DCR) is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator. For participants with a best overall response of SD, a RECIST assessment of SD must have been observed at least 6 weeks minus 1 week (at least 35 study days) following the randomization.
  The adjusted disease control rate was calculated using a logistic regression stratified by race (Chinese/Asian vs. Non-Chinese/Asian vs. Non-Asian), WHO performance status (0 vs. 1), and method used for tissue testing (central vs. local).
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Percent of Participants | 96.22 [93.14 to 97.95] | 95.02 [91.52 to 97.12]
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.4483, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.63 to 2.81] — An odds ratio greater than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

15. Secondary Outcome: Progression Free Survival 2 (PFS2) (Randomized Component)
Description: Progression Free Survival 2 is defined as the time from the date of randomization to the earliest of the progression events subsequent to that used for the primary Progression Free Survival (PFS), or death in absence of a first or second progression. The second progression event must have occurred after subsequent treatment administered after the initial progression free survival event. Any participant that was lost to follow-up, withdrew consent or discontinued for other reasons at the time of the analysis were censored at the last evaluable progression assessment. Median second progression free survival (months) calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months | 30.6 [29.0 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 27.8 [26.0 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0132, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.52 to 0.93] — A hazard ratio less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

16. Secondary Outcome: Time to First Subsequent Therapy (TFST) or Death (Randomized Component)
Description: Time to first subsequent therapy (TFST) or death is defined as the time from the date of randomization to the earlier of the date of anti- cancer therapy start date following IP discontinuation or death. Any patient not known to have had a subsequent therapy or not known to have died at the time of the analysis were censored at the last known time to have not received subsequent therapy; i.e., the last follow-up visit where this was confirmed. Median time to first subsequent therapy or death calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months | 30.7 [27.3 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 25.4 [22.8 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0159, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.56 to 0.94] — A hazard ratio less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

17. Secondary Outcome: Time to Second Subsequent Therapy (TSST) or Death (Randomized Component)
Description: Time to second subsequent therapy (TSST) or death is defined as the time from the date of randomization to the earlier of the date of second subsequent anti-cancer therapy start date following IP discontinuation or death. Any patient not known to have died at the time of the analysis and not known to have had a second subsequent therapy will be censored at the last known time to have not received second subsequent therapy, i.e., the last follow-up visit where this was confirmed. If a patient terminated the study for reason other than death before second subsequent therapy, these patients will be censored at the earliest of their last known to be alive and termination dates. Median time to second subsequent therapy or death calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months | NA [NA to NA] — Median, Lower Limit and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | 33.2 [28.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0157, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.51 to 0.93] — A hazard ratio less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

18. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Items (EORTC QLQ-C30) (Randomized Component)
Description: QLQ-C30 has 30 questions and scores range from 0-100 after a linear transformation. Questions are combined to produce symptom scales, individual symptom items, functional scales, and global health status (GHS)/quality of life (QoL).
  Positive change from baseline scores on the GHS/QoL and functioning scales indicate improvement on health status/function, and negative change scores on symptom scales/items represent less symptom severity/improvement on symptom status.
  The score values calculated by averaging across patients overall mean across all visits. The analysis was performed using a MMRM analysis on the change from baseline in the score at each visit, including subject (random effect), treatment, visit (fixed effect & repeated measure) and treatment by visit interaction as explanatory variables, with the baseline score as a covariate along with the baseline score by assessment interaction.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 253 | 253
Scores on a Scale
  Functional Scale: Physical Functioning Score (Change from Baseline) | 2.37 [0.70 to 4.04] | 6.74 [5.04 to 8.43]
  Symptom Scale: Fatigue Score (Change from Baseline) | -0.03 [-1.91 to 1.84] | -6.31 [-8.22 to -4.40]
  Individual Symptom Item: Appetite Loss Score (Change from Baseline) | 2.87 [0.82 to 4.92] | -4.58 [-6.67 to -2.48]
  Global Health Status/Quality of Life Score (Change from Baseline) | 3.32 [1.67 to 4.98] | 7.38 [5.70 to 9.07]

19. Secondary Outcome: Median Time to Deterioration in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Items (EORTC QLQ-C30) (Randomized Component)
Description: The EORTC QLQ-C30 consists of 30 questions that are combined to produce 3 symptom scales (fatigue, pain, and nausea/vomiting), 5 individual symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea), 5 functional scales (physical, role, cognitive, emotional, and social), and a global measure of health status/QoL. Scores range from 0-100 after a linear transformation.
  Time to deterioration (TTD) is defined as the time from randomization until the date of the first clinically meaningful worsening (a change in the score from baseline of ≥10) that is confirmed at a subsequent assessment or death in the absence of a clinically meaningful symptom, function, or global health status/QoL worsening, regardless of whether the patient withdraws from study treatment or receives another anticancer therapy prior to symptom, function or GHS/QoL deterioration. The median TTD was calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months
  Median TTD for Physical Functioning Scale (months) | 25.5 [17.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | NA [29.6 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Role Functioning Scale (months) | 13.1 [8.9 to 22.8] | 21.9 [18.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Cognitive Functioning Scale (months) | 15.7 [10.1 to 21.5] | 20.0 [15.4 to 25.5]
  Median TTD for Emotional Functioning Scale (months) | 29.6 [25.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | NA [NA to NA] — Median TTD, Lower Limit and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Social Functioning Scale (months) | 19.3 [11.7 to 27.8] | 28.4 [20.6 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Fatigue Symptom Scale (months) | 5.9 [2.6 to 11.8] | 20.0 [13.8 to 28.4]
  Median TTD for Pain Symptom Scale (months) | 28.0 [21.5 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 24.6 [20.0 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Nausea/Vomiting Symptom Scale (months) | 20.5 [13.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 30.5 [23.4 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Dyspnea Symptom Item (months) | NA [25.8 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | NA [21.9 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Insomnia Symptom Item (months) | NA [27.7 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | NA [23.4 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Appetite Loss Symptom Item (months) | 10.1 [5.1 to 23.0] | 28.4 [21.0 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Constipation Symptom Item (months) | 21.7 [15.9 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | NA [23.8 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Diarrhea Symptom Item (months) | 7.8 [4.4 to 11.9] | 7.7 [4.6 to 16.9]
  Median TTD for Global Health Status/Quality of Life (months) | 25.8 [20.1 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | NA [24.6 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.

20. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 Items (EORTC QLQ-LC13) (Randomized Component)
Description: EORTC QLQ-LC13 has 13 questions and scores range from 0-100 after a linear transformation. Questions assess cough, hemoptysis, dyspnea, site specific pain, sore mouth, dysphagia, peripheral neuropathy, and alopecia and pain medication. While the QLQ-LC13 includes more scales, only the Coughing, Pain in chest, and Dyspnea subscale scores were analyzed for this endpoint.
  Negative change from baseline scores indicates less symptom severity, and thus improvement on health status.
  The score values calculated by averaging across patients overall mean across all visits. The analysis was performed using a MMRM analysis on the change from baseline in the score at each visit, including subject (as a random effect), treatment, visit (as fixed effect and repeated measure) and treatment by visit interaction as explanatory variables, with the baseline score as a covariate along with the baseline score by assessment interaction.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, includes all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 253 | 251
Scores on a Scale
  Coughing Score (Change from Baseline) | -13.23 [-14.85 to -11.62] | -11.19 [-12.83 to -9.55]
  Pain in Chest Score (Change from Baseline) | -6.33 [-7.66 to -4.99] | -6.61 [-7.98 to -5.25]
  Dyspnea Score (Change from Baseline) | -3.09 [-4.70 to -1.49] | -5.67 [-7.30 to -4.04]

21. Secondary Outcome: Time to Deterioration in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 Items (EORTC QLQ-LC13) (Randomized Component)
Description: EORTC QLQ-LC13 has 13 questions and scores range from 0-100 after a linear transformation. Questions assess cough, hemoptysis, dyspnea, site specific pain, sore mouth, dysphagia, peripheral neuropathy, and alopecia and pain medication.
  Time to deterioration (TTD) is defined as the time from randomization until the date of the first clinically meaningful worsening (a change in the score from baseline of ≥10) that is confirmed at a subsequent assessment or death in the absence of a clinically meaningful symptom, function, or global health status/QoL worsening, regardless of whether the patient withdraws from study treatment or receives another anticancer therapy prior to symptom, function or GHS/QoL deterioration. The median TTD was calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Full Analysis Set, all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 279 | 278
Months
  Median TTD for Coughing Subscale (months) | NA [30.4 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | 24.7 [21.3 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Haemoptysis Subscale (months) | NA [NA to NA] — Median TTD, Lower Limit and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | NA [NA to NA] — Median TTD, Lower Limit and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Dysphagia Subscale (months) | 25.6 [20.8 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | NA [23.4 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Pain in arm or shoulder Subscale (months) | 25.2 [20.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 23.8 [18.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Pain in other parts Subscale (months) | 23.0 [15.7 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation. | 21.3 [18.2 to NA] — Upper Limit for the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.
  Median TTD for Pain in Chest Subscale (months) | NA [25.7 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off. | NA [25.2 to NA] — Median TTD and Upper Limit for the 95% confidence interval were not estimated due to the small number of participants with events at data cut off.
  Median TTD for Sore mouth Subscale (months) | 4.3 [2.1 to 7.0] | 5.8 [4.1 to 9.7]
  Median TTD for Dyspnea Subscale (months) | 9.0 [5.6 to 13.1] | 19.4 [13.7 to 24.6]
  Median TTD for Peripheral neuropathy Subscale (months) | 11.3 [7.1 to 15.7] | 15.1 [9.7 to 18.2]
  Median TTD for Alopecia Subscale (months) | 3.4 [2.8 to 4.3] | 8.9 [5.7 to 18.2]

22. Secondary Outcome: Concordance of Epidermal Growth Factor Receptor (EGFR) Mutation Status Between the Local EGFR Mutation Test and the Central Cobas® EGFR Mutation Test v2 Results: Exon 19 Deletion (Randomized Component)
Description: Comparing the local EGFR mutation test result used for patient selection with the retrospective central cobas® EGFR Mutation Test v2 results in participants with EXON 19 Deletion, excluding invalid results.
  Since this endpoint uses pre-randomization data to compare results from a central vs. local lab, randomized component treatment arms were combined for analysis.
Time Frame: Screening/Baseline
Population: Participants with a valid local and central test result.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Randomized Participants: All subjects from both randomized treatment arms: AZD9291 + Chemo and AZD9291
Arm/Group | Overall Randomized Participants
Number analyzed (Participants) | 254
Participants
  Local Laboratory Test = Negative, Cobas Central Test = Negative | 98
  Local Laboratory Test = Negative, Cobas Central Test = Positive | 0
  Local Laboratory Test = Positive, Cobas Central Test = Negative | 2
  Local Laboratory Test = Positive, Cobas Central Test = Positive | 154

23. Secondary Outcome: Concordance of Epidermal Growth Factor Receptor (EGFR) Mutation Status Between the Local EGFR Mutation Test and the Central Cobas® EGFR Mutation Test v2 Results: L858R (Randomized Component)
Description: Comparing the local EGFR mutation test result used for patient selection with the retrospective central cobas® EGFR Mutation Test v2 results in participants with L858R, excluding invalid results.
  Since this endpoint uses pre-randomization data to compare results from a central vs. local lab, randomized component treatment arms were combined for analysis.
Time Frame: Screening/Baseline
Population: Participants with a valid local and central test result.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Randomized Participants
Number analyzed (Participants) | 247
Participants
  Local Laboratory Test = Negative, Cobas Central Test = Negative | 145
  Local Laboratory Test = Negative, Cobas Central Test = Positive | 0
  Local Laboratory Test = Positive, Cobas Central Test = Negative | 6
  Local Laboratory Test = Positive, Cobas Central Test = Positive | 96

24. Secondary Outcome: Progression-free Survival (PFS) by Investigator by Plasma Epidermal Growth Factor Receptor Mutation Status: Exon 19 Deletion - Participants With an Event (Randomized Component)
Description: PFS is defined as the time from randomization until an event. An event is defined as the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the subject withdraws from study treatment or receives another anti-cancer therapy prior to progression.
  Subgroup analysis was performed using a Cox proportional hazards model including treatment, subgroup and a treatment-by subgroup interaction term.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Subgroup of Full Analysis Set, includes all randomized participants with Exon 19 Deletion EGFR mutation.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 172 | 169
Participants | 65 | 94
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; Subgroup analysis was performed using a Cox proportional hazards model including treatment, subgroup and a treatment-by subgroup interaction term; Test type: Superiority; Cox proportional hazards model; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.44 to 0.83] — A hazard ratio less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

25. Secondary Outcome: Progression-free Survival (PFS) by Investigator by Plasma Epidermal Growth Factor Receptor Mutation Status: L858R - Participants With an Event (Randomized Component)
Description: as for outcome 24
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: Subgroup of Full Analysis Set, includes all randomized participants with L858R EGFR mutation.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 106 | 107
Participants | 55 | 70
Statistical Analysis 1: Comparison: Randomized: AZD9291 + Chemo vs Randomized: AZD9291; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.44 to 0.90] — A hazard ratio less than 1 favors the Osimertinib (AZD9291) + Chemo treatment arm

26. Secondary Outcome: Plasma Concentration of Osimertinib When Given With or Without Chemotherapy (Randomized Component)
Description: An analysis will be performed to assess whether the plasma concentration of osimertinib is affected when given with or without chemotherapy. Samples were collected pre-dose and 1-hour post-dose on day 22 and day 106; on day 43 samples were collected pre-dose and 1-, 2-, 4-, and 6-hours post-dose.
Time Frame: Pre-dose and 1-hour post-dose on Day 22; pre-dose, 1-, 2-, 4-, and 6-hours post-dose on Day 43; pre-dose and 1-hour post-dose on Day 106.
Population: Pharmacokinetic Analysis Set, includes all randomized participants that received at least 1 dose of study treatment, have at least 1 measurable PK concentration and no missing doses 7 days prior to the PK sample, without any protocol deviation that affects PK, supported by the relevant date and time of this sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 244 | 263
nM
  Day 22, pre-dose: number analyzed (Participants) | 217 | 252
  Day 22, pre-dose | 430.6 (81.81) | 470.1 (46.33)
  Day 22, 1-hour post-dose: number analyzed (Participants) | 221 | 254
  Day 22, 1-hour post-dose | 430.1 (77.16) | 486.8 (46.23)
  Day 43, pre-dose: number analyzed (Participants) | 206 | 252
  Day 43, pre-dose | 401.0 (71.08) | 404.1 (53.67)
  Day 43, 1-hour post-dose: number analyzed (Participants) | 208 | 252
  Day 43, 1-hour post-dose | 401.6 (69.97) | 425.4 (54.48)
  Day 43, 2-hours post-dose: number analyzed (Participants) | 195 | 239
  Day 43, 2-hours post-dose | 457.0 (60.85) | 475.4 (52.81)
  Day 43, 4-hours post-dose: number analyzed (Participants) | 192 | 237
  Day 43, 4-hours post-dose | 525.8 (55.41) | 546.8 (46.75)
  Day 43, 6-hours post-dose: number analyzed (Participants) | 187 | 237
  Day 43, 6-hours post-dose | 544.3 (53.51) | 549.8 (45.28)
  Day 106, pre-dose: number analyzed (Participants) | 149 | 227
  Day 106, pre-dose | 393.7 (59.73) | 372.0 (53.87)
  Day 106, 1-hour post-dose: number analyzed (Participants) | 148 | 223
  Day 106, 1-hour post-dose | 407.6 (60.12) | 380.3 (54.56)

27. Secondary Outcome: Plasma Concentration of Metabolite AZ5104 When Osimertinib is Given With or Without Chemotherapy (Randomized Component)
Description: An analysis will be performed to assess whether the plasma concentration of metabolite AZ5104 is affected when given with or without chemotherapy. Samples were collected pre-dose and 1-hour post-dose on day 22 and day 106; on day 43 samples were collected pre-dose and 1-, 2-, 4-, and 6-hours post-dose.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 244 | 263
nM
  Day 22, pre-dose: number analyzed (Participants) | 217 | 252
  Day 22, pre-dose | 51.74 (82.11) | 52.42 (56.28)
  Day 22, 1-hour post-dose: number analyzed (Participants) | 221 | 254
  Day 22, 1-hour post-dose | 49.56 (81.57) | 52.78 (56.56)
  Day 43, pre-dose: number analyzed (Participants) | 206 | 252
  Day 43, pre-dose | 47.77 (80.80) | 43.89 (61.54)
  Day 43, 1-hour post-dose: number analyzed (Participants) | 208 | 252
  Day 43, 1-hour post-dose | 46.48 (80.00) | 44.89 (60.66)
  Day 43, 2-hour post-dose: number analyzed (Participants) | 195 | 239
  Day 43, 2-hour post-dose | 49.19 (71.52) | 47.14 (56.20)
  Day 43, 4-hour post-dose: number analyzed (Participants) | 192 | 237
  Day 43, 4-hour post-dose | 52.44 (67.61) | 50.92 (54.33)
  Day 43, 6-hour post-dose: number analyzed (Participants) | 187 | 237
  Day 43, 6-hour post-dose | 53.04 (65.94) | 50.89 (53.01)
  Day 106, pre-dose: number analyzed (Participants) | 150 | 227
  Day 106, pre-dose | 47.33 (64.86) | 41.09 (57.71)
  Day 106, 1-hour post-dose: number analyzed (Participants) | 148 | 223
  Day 106, 1-hour post-dose | 47.17 (65.49) | 41.30 (57.60)

28. Secondary Outcome: Mean Cmin,ss and Mean Cmax,ss of Osimertinib (Randomized Component)
Description: Cmin,ss is the minimum plasma concentration of Osimertinib at steady state. Cmax,ss is the maximum plasma concentration of Osimertinib at steady state.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 179 | 233
nmol/L
  Cmin,ss | 392.5 (50.45) | 397.2 (40.39)
  Cmax,ss | 587.5 (46.37) | 593.4 (37.26)

29. Secondary Outcome: Mean Cmin,ss and Mean Cmax,ss of AZ5104 (Randomized Component)
Description: Cmin,ss is the minimum plasma concentration of AZ5104 at steady state. Cmax,ss is the maximum plasma concentration of AZ5104 at steady state.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 179 | 233
nmol/L
  Cmin,ss | 45.34 (59.51) | 42.70 (49.42)
  Cmax,ss | 59.07 (59.80) | 55.59 (46.26)

30. Secondary Outcome: Mean AUCss of Osimertinib (Randomized Component)
Description: AUCss is the area under the plasma concentration-time curve over a doing interval at a stead state.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 176 | 233
h*nmol/L | 11840 (45.45) | 11790 (37.37)

31. Secondary Outcome: Mean AUCss of AZ5104 (Randomized Component)
Description: AUCss is the area under the plasma concentration-time curve over a doing interval at a stead state.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 176 | 233
h*nmol/L | 1277 (54.72) | 1177 (47.11)

32. Secondary Outcome: Mean CLss/F of Osimertinib (Randomized Component)
Description: CLss/F is the apparent plasma clearance at steady state.
Time Frame: Up to approximately 33 months after the first patient is randomized.
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Randomized: AZD9291 + Chemo | Randomized: AZD9291
Number analyzed (Participants) | 176 | 233
L/h | 13.52 (45.45) | 13.58 (37.37)

ADVERSE EVENTS:
Time Frame: Includes treatment emergent adverse events with onset date on or after the date of first dose and up to and including 28 days following discontinuation of treatment but prior to the start of a new anti-cancer therapy. For the Safety Run-In treatment arms, this was up to 45 months, or the data cut-off. For the Randomized treatment arms, this was up to 33 months, or the data cut-off.
Description: All AE data is based off of the Safety Analysis Set, which includes all patients who received at least 1 dose of study treatment. The All-Cause Mortality section is based off of all subjects who were assigned a study treatment in either the Safety Run-In or Randomized Treatment Arms.
Arm/Group | Safety Run-In: AZD9291 + Carboplatin + Pemetrexed | Safety Run-In: AZD9291 + Cisplatin + Pemetrexed | Randomized: AZD9291 + Chemo | Randomized: AZD9291
All-Cause Mortality (participants affected / at risk) | 6/15 | 3/15 | 71/279 | 78/278
Serious Adverse Events (participants affected / at risk) | 5/15 | 6/15 | 104/276 | 53/275
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15 | 273/276 | 258/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In: AZD9291 + Carboplatin + Pemetrexed (N=15) | Safety Run-In: AZD9291 + Cisplatin + Pemetrexed (N=15) | Randomized: AZD9291 + Chemo (N=276) | Randomized: AZD9291 (N=275)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 9 (11) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to vaccine (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 7 (8) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 7 (7) | 6 (6)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (8) | 0 (0)
Endocarditis noninfective (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 6 (8) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Otolithiasis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (6) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In: AZD9291 + Carboplatin + Pemetrexed (N=15) | Safety Run-In: AZD9291 + Cisplatin + Pemetrexed (N=15) | Randomized: AZD9291 + Chemo (N=276) | Randomized: AZD9291 (N=275)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 16 (18) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (10) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 12 (16) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 20 (22) | 7 (8)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 9 (16) | 4 (5) | 81 (95) | 28 (30)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 7 (8) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 6 (6) | 118 (225) | 112 (160)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 15 (16) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 12 (13) | 6 (6)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 67 (181) | 9 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 21 (23) | 7 (7)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (2) | 1 (1) | 18 (29) | 10 (20)
Nausea (Gastrointestinal disorders) | 3 (7) | 9 (20) | 117 (187) | 28 (33)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 3 (3) | 51 (94) | 12 (15)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (13) | 4 (6) | 68 (94) | 50 (61)
Vomiting (Gastrointestinal disorders) | 3 (5) | 0 (0) | 72 (108) | 17 (20)
Asthenia (General disorders) | 1 (1) | 0 (0) | 26 (41) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (5) | 123 (210) | 22 (26)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (4) | 5 (5)
Face oedema (General disorders) | 1 (1) | 1 (1) | 10 (10) | 2 (2)
Fatigue (General disorders) | 2 (2) | 2 (2) | 76 (129) | 25 (28)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 7 (8) | 6 (11)
Malaise (General disorders) | 0 (0) | 2 (2) | 19 (24) | 3 (3)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 24 (29) | 14 (16)
Oedema (General disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 5 (5) | 42 (50) | 12 (12)
Pain (General disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 30 (36) | 15 (19)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (4) | 3 (4)
COVID-19 (Infections and infestations) | 3 (3) | 5 (5) | 50 (52) | 37 (38)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 16 (18) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 6 (9)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 7 (7) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 8 (8)
Oral candidiasis (Infections and infestations) | 1 (2) | 1 (1) | 5 (5) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 9 (9) | 4 (6) | 65 (74) | 73 (100)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 8 (8) | 10 (12)
Purulence (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3) | 16 (20) | 9 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 34 (55) | 27 (39)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 7 (7) | 5 (7)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 56 (108) | 21 (27)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 48 (111) | 13 (20)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 9 (12) | 7 (7)
Blood creatinine increased (Investigations) | 0 (0) | 3 (4) | 45 (67) | 12 (19)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 13 (22) | 11 (14)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 13 (14) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 17 (17) | 9 (10)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 24 (36) | 23 (33)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 17 (28) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 62 (259) | 16 (27)
Platelet count decreased (Investigations) | 3 (3) | 1 (1) | 51 (117) | 19 (31)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 32 (34) | 22 (25)
Weight increased (Investigations) | 0 (0) | 2 (5) | 13 (17) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 44 (218) | 18 (37)
Acquired mixed hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 1 (1) | 81 (116) | 25 (28)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 12 (24) | 11 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (7) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 17 (29) | 13 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 18 (24) | 12 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 18 (24) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 16 (27) | 12 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 27 (29) | 32 (38)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 23 (23) | 26 (28)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 9 (9) | 15 (15)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 11 (12) | 15 (16)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 8 (8) | 14 (16)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 9 (9) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 8 (9) | 16 (24)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 5 (6) | 4 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 32 (38) | 16 (17)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0) | 17 (17) | 11 (13)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 26 (28) | 26 (35)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 9 (11) | 5 (7)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 13 (13) | 6 (7)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1) | 34 (36) | 18 (18)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 12 (13) | 7 (8)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 31 (35) | 29 (35)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 15 (15) | 15 (17)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 20 (28) | 18 (21)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (5) | 11 (13) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 4 (5) | 4 (4)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 18 (19) | 7 (7)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 6 (6) | 2 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 8 (9) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 24 (24) | 15 (15)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 7 (9) | 7 (7)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (5) | 37 (47) | 36 (51)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 50 (57) | 66 (70)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (13) | 2 (2) | 4 (5)
Follicular disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 10 (11)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 15 (18) | 9 (9)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 22 (28) | 31 (39)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6) | 77 (98) | 57 (75)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 18 (24) | 19 (21)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 34 (132) | 11 (17)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 7 (7) | 7 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 7 (8) | 3 (3)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 18 (21) | 15 (17)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (2) | 1 (4) | 12 (12) | 8 (8)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to submit all manuscripts or abstracts to the sponsor before submission for publication or presentation at scientific meetings to allow the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04035486/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT04035486/SAP_002.pdf